CLINICAL TRIAL: NCT03383978
Title: Multicenter, Open Label, Phase I Study of Intracranial Injection of NK-92/5.28.z Cells in Patients With Recurrent HER2-positive Glioblastoma
Brief Title: Intracranial Injection of NK-92/5.28.z Cells in Combination With Intravenous Ezabenlimab in Patients With Recurrent HER2-positive Glioblastoma
Acronym: CAR2BRAIN
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: DRK Blutspendedienst Baden-Württemberg-Hessen gGmbH (Unknown); Georg-Speyer-Haus (Unknown); LOEWE Center Frankfurt Cancer Institute (Unknown); German Cancer Research Center (Other)
Responsible Party: Principal Investigator, Michael Burger, Principal Investigator, Johann Wolfgang Goethe University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2016-000225-39
Record Dates: First submitted 2017-11-30; First posted 2017-12-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NK-92/5.28.z + Ezabenlimab (Experimental): Intracranial application of NK-92/5.28.z, 1x10E7-1x10E8; intravenous infusion of Ezabenlimab 240mg q 3 weeks
  Interventions: Biological: NK-92/5.28.z; Drug: Ezabenlimab

INTERVENTIONS:
Biological: NK-92/5.28.z — Intracranial application of NK-92/5.28.z, 1x10E7-1x10E8
Drug: Ezabenlimab — Intravenous infusion of Ezabenlimab 240mg q 3 weeks

SUMMARY:
The main objective of this clinical study is to evaluate the safety and tolerability of NK-92/5.28.z and to determine the maximum tolerated dose or maximum feasible dose (MFD). Recommended phase 2 doses both for intraoperative injections only (RP2Diio) and repetitive injections (RP2Dri) will be determined. Frequent side effects and target organs of toxicity and their severity, duration and reversibility will be determined. Furthermore, pharmacokinetics and pharmacodynamics will be examined. In addition, potential signs of anti-tumor activity of NK-92/5.28.z cells will be analyzed. In the separate "CAR2BRAIN-Check" cohort, combination therapy of NK-92/5.28.z with the anti-PD-1 antibody Ezabenlimab (BI 754091) will be tested.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent or refractory HER2-positive glioblastoma or its variant gliosarcoma in which relapse surgery (partial or total) or a biopsy (biopsy only for the "CAR2BRAIN-Check" cohort) is being planned. Those patients with planned biopsy may be included into the "CAR2BRAIN-Check" cohort, if all of the following conditions apply:

   * Biopsy is necessary (as determined by the treating physician) to rule out the differential diagnosis of pseudoprogression prior to relapse surgery.
   * Suspected tumor relapse is located in the wall of an already existing resection cavity.
   * This resection cavity has a volume of at least 2.5 ml or is connected to a ventricle or has a broad connection to the surface of the brain.
   * Patients must be candidates for relapse surgery, which must be postponable for four weeks.
2. Prior therapy must include the standard of care for glioblastoma (radiotherapy and alkylating chemotherapy, or at least a part thereof if the therapy was terminated prematurely due to therapy failure or poor tolerance). For patients with non-methylated MGMT-Promotor, prior alkylating chemotherapy is dispensable.
3. Age ≥ 18 years
4. Life expectancy ≥ 3 months
5. Bilirubin ≤ 3x normal, AST ≤ 5x normal, ALT ≤ 5x normal, serum creatinine ≤ 2x upper limit of normal for age, leukocyte count ≥ 3/nl, thrombocyte count ≥ 100/nl and Hb ≥ 8.0 g/dl
6. Blood oxygenation of ≥ 90% as measured by pulse oximetry on room air
7. Women must have a negative serum pregnancy test within 72h prior to the start of the first NK-92/5.28.z cell injection.
8. Sexually active patients must be willing to utilize effective birth control methods throughout the study and for 24 weeks after the last NK-92/5.28.z cell injection. This includes two different forms of effective contraception (e.g. hormonal contraceptive and condom, IUD/IUS and condom) or sterilization.
9. Patients should have been off other antineoplastic therapy for two weeks prior to entry in this study. Temozolomide will be allowed up to 48h preinjection. At the time of inclusion, dexamethasone up to a total dose of 4 mg per day will be allowed if medically indicated.
10. Informed consent explained to and signed by patient; patient given copy of informed consent.
11. Karnofsky performance score of ≥ 70%

Exclusion criteria:

1. Anti-angiogenic therapy e.g. with bevacizumab in the last four weeks prior to study entry
2. Previous anti-PD-1 or anti-PD-L1 directed checkpoint inhibitor therapy (only "CAR2BRAIN-Check" cohort)
3. Coagulation disorder (INR>1.4 or PTT>50sec) or anticoagulation in therapeutic dosage
4. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. However, patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study.
5. Patients with Type I diabetes mellitus not on a stable dose of insulin regimen
6. Psoriatic arthritis (however, patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only are permitted provided that they meet all of the following conditions:

   * Rash must cover less than 10% of body surface area
   * Disease is well controlled at baseline and only requiring low potency topical steroids
   * No acute exacerbations of underlying condition within the previous 12 months (not requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high potency or oral steroids))
7. Patients with clinical or laboratory signs for immunodeficiency or under immunosuppressive medication other than corticosteroids
8. Severe intercurrent infection
9. Known HIV, HBV (defined by detection of HBsAg) or HCV positivity (defined by detection of HCV-IgG)
10. Chronic heart failure NYHA ≥III
11. Patients with a prior solid organ transplantation or allogenic haematopoietic stem cell transplantation
12. Patients unable to undergo MRI
13. Pregnancy or breastfeeding
14. Drug or alcohol abuse
15. Severe psychiatric disorder which might interfere with the study treatment or examination
16. Simultaneous participation in another interventional clinical trial. If a subject participated in a trial testing another IMP, such IMP should have been terminated at least 30 days before inclusion of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03. | 24 weeks
Maximum tolerated dose (MTD) or maximum feasible dose (MFD) for NK-92/5.28.z | 24 weeks
Period of detectability of NK-92/5.28.z cells in blood and cerebrospinal fluid (CSF) during the first 24 weeks after NK-92/5.28.z application with qPCR. | 24 weeks
  qPCR detection of NK-92/5.28.z in blood or CSF
Cytokine profile in the blood and the cerebrospinal fluid. | 24 weeks

SECONDARY OUTCOMES:
NK-92- and/or CAR 5.28.z-directed immune response. | 24 weeks
Objective response rate. | 24 weeks
Progression-free survival. | 24 weeks
Overall survival. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Burger, PD Dr. med., Principal Investigator — Johann W. Goethe University Hospital, Frankfurt am Main, Germany
Locations (4):
- Germany (4):
  - Neurochirurgische Klinik, Universitätsmedizin Mannheim, Mannheim, Baden-Wurttemberg
  - Neurochirurgische Klinik, Universitätsmedizin Mainz, Mainz, Rhineland-Palatinate
  - Johann W. Goethe University Hospital, Department of Neurosurgery, Frankfurt
  - Johann W. Goethe University Hospital, Senckenberg Institute of Neurooncology, Frankfurt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor homepage — https://www.kgu.de/einrichtungen/kliniken/zentrum-der-neurologie-und-neurochirurgie/dr-senckenbergisches-institut-fuer-neuroonkologie/unser-institut/